CLINICAL TRIAL: NCT01911494
Title: The CLIP (Community Level Interventions for Pre-eclampsia) Cluster Randomized Controlled Trial
Brief Title: Community Level Interventions for Pre-eclampsia
Acronym: CLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Olabisi Onabanjo University (Other); Centro de Investigacao em Saude de Manhica (Other); Aga Khan University (Other); Jawaharlal Nehru Medical College (Other)
Responsible Party: Principal Investigator, Peter von Dadelszen, Study Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H12-03497; F12-01593 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2013-06-28; First posted 2013-07-30 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Pre-eclampsia; Hypertension, Pregnancy Induced
Keywords: cluster randomized controlled trial; pre-eclampsia; eclampsia; maternal mortality
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Eclampsia; Maternal Death | interventions — Magnesium Sulfate; Methyldopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The CLIP intervention consists of (i) community engagement including community leaders, the women of the communities themselves, and their mothers, husbands, and mothers-in-law, regarding pre-eclampsia, its origins, symptoms, signs, and potential consequences, pre-permissions for maternal transport, and fundraising activities around transport and treatment costs; (ii) provision of HDP oriented antenatal care through CLIP visits and use of CLIP "PIERS on the Move" mHealth tool (for risk stratification), and (iii) use of the CLIP package for women with a CLIP 'trigger' (i.e., oral antihypertensive therapy (methyldopa) when indicated, intramuscular (i.m.) magnesium sulfate when indicated; and appropriate referral to an CEmOC facility when indicated)
  Interventions: Behavioral: Community Engagement; Device: PIERS on the Move mHealth decision aid; Drug: Magnesium Sulfate; Drug: Methyldopa
- Control (No Intervention): Current standard of antenatal care

INTERVENTIONS:
Behavioral: Community Engagement — The primary objective of the community engagement activities in CLIP will be to create awareness and action around the prevention of maternal morbidity and mortality due to pre-eclampsia/eclampsia. Community engagement involves the collective action of individuals, families, religious leaders, policy makers,
  Arms: Intervention
Device: PIERS on the Move mHealth decision aid — This mHealth application is to be used by community health workers in intervention clusters to guide collection of relevant clinical data during antenatal visits. This clinical data is used to generate a risk estimate for any women with hypertension based on the miniPIERS (Pre-eclampsia Integrated Estimate of Risk) clinical risk prediction model. This risk estimate in combination with other pre-defined treatment triggers (severe hypertension (>160mmHg systolic) or proteinuria (>3+ dipstick); absence of fetal movements for greater than 12 hours; signs of recent stroke of seizure) are collected in the app and based on this data recommendations for care of the woman are provided.
  Other Names: CLIP mHealth tool
  Arms: Intervention
Drug: Magnesium Sulfate — Women identified in intervention clusters by the community health worker during a study visit as being at high risk of- or having recently experienced- an eclamptic seizure will be given 10 g intramuscular magnesium sulfate prior to transfer to a nearby facility for further care.
  Other Names: MgSO4
  Arms: Intervention
Drug: Methyldopa — Women identified in intervention clusters as having severe hypertension (systolic greater than 160 mmHg) by the community health worker during a study visit will be given 750 mg of oral methyldopa prior to transfer to a nearby facility for further care.
  Other Names: Aldomet
  Arms: Intervention

SUMMARY:
This project is being undertaken to test the hypothesis that implementing a community based package of care for women with hypertensive disorders of pregnancy will result in overall improvement in maternal and neonatal outcomes. This is based on the premise that there are three main modifiable reasons why women (and their fetuses/newborns) die due to pregnancy complications: 1) delays by the woman herself in recognizing the seriousness of her condition; 2) delays in her being assessed and then transported to a center capable of providing effective and life-saving interventions; and 3) delays in the health facility in providing those interventions. The treatments for pre-eclampsia that are poorly accessed in LMIC are 1) magnesium sulfate (MgSO4) for prevention and treatment of the grand mal seizures of eclampsia; 2) oral antihypertensive medication to lower maternal BP to reduce the risk of stroke.

The CLIP pilot and definitive cRCT will investigate whether the community level intervention including implementation of the CLIP package (oral antihypertensive therapy when indicated, intramuscular (i.m.) MgSO4 when indicated; and appropriate referral to an CEmOC facility when indicated) of care will reduce the incidence of all-cause maternal morbidity and mortality.

DETAILED DESCRIPTION:
We have designed a two-phased community (including PHC-level) cRCT encompassing both rural and urban settings to be fully powered in each of:

* Ogun State, Nigeria
* Maputo and Gaza Province, Mozambique
* Hyderabad and Matiari districts in Sindh Province, Pakistan.
* Belgaum and Bagalkot districts in Karnataka State, India The trial will be phased from the Pilot CLIP trial to Definitive CLIP trial on the basis of a satisfactory rate of use (≥50%) of the CLIP 'package of care' in appropriate women in all countries but Mozambique. Mozambique will be unique in that they will rely on an extended period of feasibility to pilot test all Trial systems and tools before directly beginning a definitive trial. Foregoing the Pilot in Mozambique was felt to be appropriate based on their experience with community-based surveillance and will ensure timelines of the trial are met within a manageable budget.

For all other countries, use of the package in the Pilot phase will be defined as appropriate referral (urgent or non-urgent) to a facility able to provide comprehensive emergency obstetric care (CEmOC) in appropriate women during the first six months of the Pilot CLIP trial.

A primary component of the CLIP intervention is antenatal risk assessment guided by the PIERS on teh Move mHealth decision aid. The CLIP version of the PIERS on the Move tool (CLIP POM) integrates the miniPIERS predictive score and a clinical data collection system into a single application. Community health workers in each country will assess women according to the visit protocol, entering clinical data into the CLIP POM mobile application. The application will provide recommendations for care according to meeting one of the trigger events listed below, as per this protocol. Triggers identified that will indicate treatment and/or transport (urgently, defined as within 4hrs) to a CEmOC facility are as follows:

1. Unconsciousness (MgSO4 if sBP ≥160 mmHg [to be reasonably sure that the unconsciousness is associated with severe pre-eclampsia and not due to obstetric sepsis], urgent transport)
2. Signs of recent stroke or seizure (methyldopa if sBP ≥160 mmHg [to ensure BP is not lowered too much], MgSO4, urgent transport)
3. Significant vaginal bleeding (MgSO4 if sBP ≥140 mmHg [presumed abruption associated with severe pre-eclampsia], urgent transport).
4. No fetal movements felt in the previous 12 hrs (urgent transport [a threshold for identifying at risk fetuses that are alive at the time of screening] 39)
5. sBP ≥160 mmHg (or dBP ≥ 110 mmHg in Nigeria only) (methyldopa, MgSO4, urgent transport [consistent with severe pre-eclampsia])
6. Heavy proteinuria (≥4+ by dipstick - predictive of stillbirth in miniPIERS cohort, urgent transport)
7. miniPIERS predicted probability ≥25% (MgSO4, urgent transport)
8. Shock index >1.7 in Nigeria only (the Shock index is a ratio of pulse/sBP; high shock index is an indication of poor prognosis in women with postpartum haemorrhage) Non-urgent transport (by non-ambulance services), meaning assessment at a CEmOC facility within 24 hours, will be advised for all women with non-severe hypertension (sBP 140-159 mmHg) who do not meet criteria for one of the above 7/8 triggers.

In Mozambique and Pakistan additional CLIP triggers based on use of the audio oximeter will also be included in the POM decision aid. As with the original miniPIERS model, the enhanced model including SpO2 uses a risk threshold of ≥25% predicted probability to identify high-risk cases. Recommendations based on the updated miniPIERS model will include treatment with MgSO4 and urgent referral. An additional independent trigger of SpO2<93% will also be used in Mozambique and Pakistan to indicate urgent referral.

In Nigeria where the updated Microlife CRADLE VSA blood pressure device is being used additional triggers will be included for severe diastolic blood pressure or severe shock index to coincide with the traffic light warning signs included in this device.

ELIGIBILITY:
Inclusion Criteria:

* all consenting pregnant women

Exclusion Criteria:

* non-pregnant

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 87500 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Maternal or Perinatal death or morbidity | within 42 days of pregnancy
  Combined outcome including any one of the following:
  1. Maternal death (number of deaths during or within 42d of pregnancy or last contact day if contact not maintained to 42d/1000 identified pregnancies); termed Maternal Death Rate.
  2. Maternal morbidity (number of women with ≥1 life-threatening complication of pregnancy (ie eclampsia, major PPH requiring surgical intervention, obstetric sepsis, stroke, etc) during or within 42d of pregnancy or last contact day if contact not maintained to 42d) / 1000 identified pregnancies
  3. Perinatal death (stillbirth [≥20+0 and/or ≥500g], early neonatal mortality [d0-7 of postnatal life] and late neonatal mortality [d8-28 of postnatal life] /1000 identified pregnancies)
  4. Neonatal morbidity (occurrence of any non-lethal morbidity (ie severe breathing difficulty, severe feeding difficulty, seizure, lethargy, coma, hypothermia, skin or umbilical stump infection, jaundice, etc) during 0-28d of postnatal life /1000 identified pregnancies)

SECONDARY OUTCOMES:
Birth preparedness and complication readiness | from 20 weeks gestation to delivery
  as measured by any three of the following: (1) arranged for transport; (2) obtained prior permission for transport should emergency arise; (3) saved money for obstetric care; (4) identified skilled birth attendant; (5) identified facility for delivery. This will evaluate the success of community engagement.
Facility births | from 20 weeks gestation to delivery
  number of women presenting for delivery in a CEmONC facility in control vs intervention clusters

OTHER OUTCOMES:
Pre-eclampsia knowledge | from 20 weeks gestation to time of delivery
Post-trial seizures | within 42 days of pregnancy
  Assessment of post-trial start eclamptic seizures in control vs intervention clusters to assess effectiveness of community dosing of magnesium sulfate
Cost-effectiveness | within 42 days of pregnancy
  Of the CLIP package against QALYs
Adverse effects | within 42 days of pregnancy
  Adverse effects of magnesium include injection site hematoma or infection, and respiratory depression
Functional disability | within 6 months of delivery
  Index measurement of functional ability, including ability to care for baby, do household chores and return to work within 6 months of delivery measured at two to four week intervals postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Peter von Dadelszen, MBChB, DPhil, Principal Investigator — University of British Columbia
Locations (4):
- Jawaharlal Nehru Medical College, Karnataka Lingayat Education University, Belagavi, Karnataka, India
- Centro de Investigacaoem Saude de Manhica (CISM), Maputo, Mozambique
- Centre for Research in Reproductive Health, Olabisi Onabanjo University, Sagamu, Ogun State, Nigeria
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Payne BA, Hutcheon JA, Ansermino JM, Hall DR, Bhutta ZA, Bhutta SZ, Biryabarema C, Grobman WA, Groen H, Haniff F, Li J, Magee LA, Merialdi M, Nakimuli A, Qu Z, Sikandar R, Sass N, Sawchuck D, Steyn DW, Widmer M, Zhou J, von Dadelszen P; miniPIERS Study Working Group. A risk prediction model for the assessment and triage of women with hypertensive disorders of pregnancy in low-resourced settings: the miniPIERS (Pre-eclampsia Integrated Estimate of RiSk) multi-country prospective cohort study. PLoS Med. 2014 Jan;11(1):e1001589. doi: 10.1371/journal.pmed.1001589. Epub 2014 Jan 21. PMID 24465185
- [Background] von Dadelszen P, Firoz T, Donnay F, Gordon R, Justus Hofmeyr G, Lalani S, Payne BA, Roberts JM, Teela KC, Vidler M, Sawchuck D, Magee LA. Preeclampsia in low and middle income countries-health services lessons learned from the PRE-EMPT (PRE-Eclampsia-Eclampsia Monitoring, Prevention and Treatment) project. J Obstet Gynaecol Can. 2012 Oct;34(10):917-926. doi: 10.1016/S1701-2163(16)35405-6. PMID 23067947
- [Background] Dunsmuir DT, Payne BA, Cloete G, Petersen CL, Gorges M, Lim J, von Dadelszen P, Dumont GA, Ansermino JM. Development of mHealth applications for pre-eclampsia triage. IEEE J Biomed Health Inform. 2014 Nov;18(6):1857-64. doi: 10.1109/JBHI.2014.2301156. PMID 25375683
- [Derived] Vidler M, Kinshella MW, Sevene E, Lewis G, von Dadelszen P, Bhutta Z; CLIP Working Group. Transitioning from the "Three Delays" to a focus on continuity of care: a qualitative analysis of maternal deaths in rural Pakistan and Mozambique. BMC Pregnancy Childbirth. 2023 Oct 23;23(1):748. doi: 10.1186/s12884-023-06055-w. PMID 37872504
- [Derived] Kavi A, Kinshella MW, Ramadurg UY, Charantimath U, Katageri GM, Karadiguddi CC, Honnungar NV, Bannale SG, Mungarwadi GI, Bone JN, Vidler M, Magee L, Mallapur A, Goudar SS, Bellad M, Derman R, von Dadelszen P, Working Group TCI. Community engagement for birth preparedness and complication readiness in the Community Level Interventions for Pre-eclampsia (CLIP) Trial in India: a mixed-method evaluation. BMJ Open. 2022 Dec 20;12(12):e060593. doi: 10.1136/bmjopen-2021-060593. PMID 36600428
- [Derived] Hoodbhoy Z, Sheikh SS, Qureshi R, Memon J, Raza F, Kinshella MW, Bone JN, Vidler M, Sharma S, Payne BA, Magee LA, von Dadelszen P, Bhutta ZA; CLIP Pakistan Working Group*. Role of community engagement in maternal health in rural Pakistan: Findings from the CLIP randomized trial. J Glob Health. 2021 Jul 17;11:04045. doi: 10.7189/jogh.11.04045. eCollection 2021. PMID 34326995
- [Derived] Bone JN, Magee LA, Singer J, Nathan H, Qureshi RN, Sacoor C, Sevene E, Shennan A, Bellad MB, Goudar SS, Mallapur AA, Munguambe K, Vidler M, Bhutta ZA, von Dadelszen P; CLIP study group. Blood pressure thresholds in pregnancy for identifying maternal and infant risk: a secondary analysis of Community-Level Interventions for Pre-eclampsia (CLIP) trial data. Lancet Glob Health. 2021 Aug;9(8):e1119-e1128. doi: 10.1016/S2214-109X(21)00219-9. Epub 2021 Jul 5. PMID 34237265
- [Derived] Bone JN, Khowaja AR, Vidler M, Payne BA, Bellad MB, Goudar SS, Mallapur AA, Munguambe K, Qureshi RN, Sacoor C, Sevene E, Frederix GWJ, Bhutta ZA, Mitton C, Magee LA, von Dadelszen P; CLIP Trials Working Group. Economic and cost-effectiveness analysis of the Community-Level Interventions for Pre-eclampsia (CLIP) trials in India, Pakistan and Mozambique. BMJ Glob Health. 2021 May;6(5):e004123. doi: 10.1136/bmjgh-2020-004123. PMID 34031134
- [Derived] Makacha L, Makanga PT, Dube YP, Bone J, Munguambe K, Katageri G, Sharma S, Vidler M, Sevene E, Ramadurg U, Charantimath U, Revankar A, von Dadelszen P. Is the closest health facility the one used in pregnancy care-seeking? A cross-sectional comparative analysis of self-reported and modelled geographical access to maternal care in Mozambique, India and Pakistan. Int J Health Geogr. 2020 Feb 3;19(1):1. doi: 10.1186/s12942-020-0197-5. PMID 32013994
- [Derived] Magee LA, Sharma S, Nathan HL, Adetoro OO, Bellad MB, Goudar S, Macuacua SE, Mallapur A, Qureshi R, Sevene E, Sotunsa J, Vala A, Lee T, Payne BA, Vidler M, Shennan AH, Bhutta ZA, von Dadelszen P; CLIP Study Group. The incidence of pregnancy hypertension in India, Pakistan, Mozambique, and Nigeria: A prospective population-level analysis. PLoS Med. 2019 Apr 12;16(4):e1002783. doi: 10.1371/journal.pmed.1002783. eCollection 2019 Apr. PMID 30978179
- [Derived] Makanga PT, Sacoor C, Schuurman N, Lee T, Vilanculo FC, Munguambe K, Boene H, Ukah UV, Vidler M, Magee LA, Sevene E, von Dadelszen P, Firoz T; CLIP Working Group. Place-specific factors associated with adverse maternal and perinatal outcomes in Southern Mozambique: a retrospective cohort study. BMJ Open. 2019 Feb 19;9(2):e024042. doi: 10.1136/bmjopen-2018-024042. PMID 30782892
- [Derived] Sharma S, Adetoro OO, Vidler M, Drebit S, Payne BA, Akeju DO, Adepoju A, Jaiyesimi E, Sotunsa J, Bhutta ZA, Magee LA, von Dadelszen P, Dada O. A process evaluation plan for assessing a complex community-based maternal health intervention in Ogun State, Nigeria. BMC Health Serv Res. 2017 Mar 28;17(1):238. doi: 10.1186/s12913-017-2124-4. PMID 28351355
- [Derived] Bellad MB, Vidler M, Honnungar NV, Mallapur A, Ramadurg U, Charanthimath U, Katageri G, Bannale S, Kavi A, Karadiguddi C, Sharma S, Lee T, Li J, Payne B, Magee L, von Dadelszen P, Derman R, Goudar SS; CLIP Working Group. Maternal and Newborn Health in Karnataka State, India: The Community Level Interventions for Pre-Eclampsia (CLIP) Trial's Baseline Study Results. PLoS One. 2017 Jan 20;12(1):e0166623. doi: 10.1371/journal.pone.0166623. eCollection 2017. PMID 28107350
- [Derived] Akeju DO, Vidler M, Sotunsa JO, Osiberu MO, Orenuga EO, Oladapo OT, Adepoju AA, Qureshi R, Sawchuck D, Adetoro OO, von Dadelszen P, Dada OA; CLIP Nigeria Feasibility Working Group. Human resource constraints and the prospect of task-sharing among community health workers for the detection of early signs of pre-eclampsia in Ogun State, Nigeria. Reprod Health. 2016 Sep 30;13(Suppl 2):111. doi: 10.1186/s12978-016-0216-y. PMID 27719681
- [Derived] Salam RA, Qureshi RN, Sheikh S, Khowaja AR, Sawchuck D, Vidler M, von Dadelszen P, Zaidi S, Bhutta Z; CLIP working group. Potential for task-sharing to Lady Health Workers for identification and emergency management of pre-eclampsia at community level in Pakistan. Reprod Health. 2016 Sep 30;13(Suppl 2):107. doi: 10.1186/s12978-016-0214-0. PMID 27719680
- [Derived] Ramadurg U, Vidler M, Charanthimath U, Katageri G, Bellad M, Mallapur A, Goudar S, Bannale S, Karadiguddi C, Sawchuck D, Qureshi R, von Dadelszen P, Derman R; Community Level Interventions for Pre-eclampsia (CLIP) India Feasibility Working Group. Community health worker knowledge and management of pre-eclampsia in rural Karnataka State, India. Reprod Health. 2016 Sep 30;13(Suppl 2):113. doi: 10.1186/s12978-016-0219-8. PMID 27719678
- [Derived] Sotunsa JO, Vidler M, Akeju DO, Osiberu MO, Orenuga EO, Oladapo OT, Qureshi R, Sawchuck D, Adetoro OO, von Dadelszen P, Dada OA; CLIP Nigeria Feasibility Working Group. Community health workers' knowledge and practice in relation to pre-eclampsia in Ogun State, Nigeria: an essential bridge to maternal survival. Reprod Health. 2016 Sep 30;13(Suppl 2):108. doi: 10.1186/s12978-016-0218-9. PMID 27719677
- [Derived] Sheikh S, Qureshi RN, Khowaja AR, Salam R, Vidler M, Sawchuck D, von Dadelszen P, Zaidi S, Bhutta Z; CLIP Working Group. Health care provider knowledge and routine management of pre-eclampsia in Pakistan. Reprod Health. 2016 Sep 30;13(Suppl 2):104. doi: 10.1186/s12978-016-0215-z. PMID 27719673
- [Derived] Vidler M, Charantimath U, Katageri G, Ramadurg U, Karadiguddi C, Sawchuck D, Qureshi R, Dharamsi S, von Dadelszen P, Derman R, Goudar S, Mallapur A, Bellad M; Community Level Interventions for Pre-eclampsia (CLIP) India Feasibility Working Group. Community perceptions of pre-eclampsia in rural Karnataka State, India: a qualitative study. Reprod Health. 2016 Jun 8;13 Suppl 1(Suppl 1):35. doi: 10.1186/s12978-016-0137-9. PMID 27358068
- [Derived] Boene H, Vidler M, Sacoor C, Nhama A, Nhacolo A, Bique C, Alonso P, Sawchuck D, Qureshi R, Macete E, Menendez C, von Dadelszen P, Sevene E, Munguambe K. Community perceptions of pre-eclampsia and eclampsia in southern Mozambique. Reprod Health. 2016 Jun 8;13 Suppl 1(Suppl 1):33. doi: 10.1186/s12978-016-0135-y. PMID 27357840
- [Derived] Akeju DO, Vidler M, Oladapo OT, Sawchuck D, Qureshi R, von Dadelszen P, Adetoro OO, Dada OA; CLIP Nigeria Feasibility Working Group. Community perceptions of pre-eclampsia and eclampsia in Ogun State, Nigeria: a qualitative study. Reprod Health. 2016 Jun 8;13 Suppl 1(Suppl 1):57. doi: 10.1186/s12978-016-0134-z. PMID 27357695
- [Derived] Khowaja AR, Qureshi RN, Sawchuck D, Oladapo OT, Adetoro OO, Orenuga EA, Bellad M, Mallapur A, Charantimath U, Sevene E, Munguambe K, Boene HE, Vidler M, Bhutta ZA, von Dadelszen P; CLIP Working Group. The feasibility of community level interventions for pre-eclampsia in South Asia and Sub-Saharan Africa: a mixed-methods design. Reprod Health. 2016 Jun 8;13 Suppl 1(Suppl 1):56. doi: 10.1186/s12978-016-0133-0. PMID 27357579
- [Derived] Munguambe K, Boene H, Vidler M, Bique C, Sawchuck D, Firoz T, Makanga PT, Qureshi R, Macete E, Menendez C, von Dadelszen P, Sevene E. Barriers and facilitators to health care seeking behaviours in pregnancy in rural communities of southern Mozambique. Reprod Health. 2016 Jun 8;13 Suppl 1(Suppl 1):31. doi: 10.1186/s12978-016-0141-0. PMID 27356968
- [Derived] Qureshi RN, Sheikh S, Khowaja AR, Hoodbhoy Z, Zaidi S, Sawchuck D, Vidler M, Bhutta ZA, von Dadeslzen P; CLIP Working Group. Health care seeking behaviours in pregnancy in rural Sindh, Pakistan: a qualitative study. Reprod Health. 2016 Jun 8;13 Suppl 1(Suppl 1):34. doi: 10.1186/s12978-016-0140-1. PMID 27356863
- [Derived] Akeju DO, Oladapo OT, Vidler M, Akinmade AA, Sawchuck D, Qureshi R, Solarin M, Adetoro OO, von Dadelszen P; CLIP Nigeria Feasibility Working Group. Determinants of health care seeking behaviour during pregnancy in Ogun State, Nigeria. Reprod Health. 2016 Jun 8;13 Suppl 1(Suppl 1):32. doi: 10.1186/s12978-016-0139-7. PMID 27356754
- [Derived] Vidler M, Ramadurg U, Charantimath U, Katageri G, Karadiguddi C, Sawchuck D, Qureshi R, Dharamsi S, Joshi A, von Dadelszen P, Derman R, Bellad M, Goudar S, Mallapur A; Community Level Interventions for Pre-eclampsia (CLIP) India Feasibility Working Group. Utilization of maternal health care services and their determinants in Karnataka State, India. Reprod Health. 2016 Jun 8;13 Suppl 1(Suppl 1):37. doi: 10.1186/s12978-016-0138-8. PMID 27356502
- [Derived] Khowaja AR, Mitton C, Bryan S, Magee LA, Bhutta ZA, von Dadelszen P. Economic evaluation of Community Level Interventions for Pre-eclampsia (CLIP) in South Asian and African countries: a study protocol. Implement Sci. 2015 May 26;10:76. doi: 10.1186/s13012-015-0266-5. PMID 26007682
- See also: CLIP trial website — https://pre-empt.bcchr.ca/treatment/clip-community-level-interventions-pre-eclampsia